CLINICAL TRIAL: NCT05928975
Title: Effects of Manual Therapy Plus Pain Neuroscience Education With Integrated Motivational Interviewing on Pain, Disability, Kinesiophobia and Catastrophizing in Individuals With Non-Specific Chronic Low Back Pain: A Randomized Clinical Trial Study
Brief Title: Manual Therapy Plus Pain Neuroscience Education With Integrated Motivational Interviewing in Individuals With Non-Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras, Principal Investigator, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-08/2022
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Non-specific Chronic Low Back pain; Manual therapy; Pain neuroscience education; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Sixty participants with non-specific chronic low back pain will be randomly assigned to three groups of 20 each. The allocation of the sample to the groups will be performed using a randomization program (https://www.randomizer.org/) by an independent researcher. The first group will receive MT and PNE with MI, the second group will receive MT alone, while participants in the control group (third group) will follow a home-based exercise program. Participants of the two intervention groups will follow a total of 10 treatment sessions over a period of 4 weeks.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MT+ PNE with MI (Experimental): Participants allocated to this group will receive 10 sessions of MT, along with 4 sessions of PNE with MI, over a period of four weeks.
  Interventions: Other: MT+ PNE with MI
- MT (Experimental): Participants allocated to this group will receive 10 sessions of MT (without PNE with MI), over a period of four weeks.
  Interventions: Other: MT
- Control (Active Comparator): Participants allocated to this group will engage in a home-based general exercise program.
  Interventions: Other: Control

INTERVENTIONS:
Other: MT+ PNE with MI — The manual therapy treatment approach entailed the management of symptoms based on the clinical judgment of the attending physiotherapist. The physiotherapist selectively employed techniques such as spinal mobilization/manipulation, soft tissue massage, supervised exercises and muscle and neural mobilization, while excluding the utilization of electrophysical modalities. The participants will receive 10 Manual Therapy sessions of 30 minutes within a period of 4 weeks.
  The pain neuroscience education program is based on previous clinical studies and available educational materials and is enhanced by motivational interviewing techniques. The program consisted of 4 individualized educational sessions, each lasting 30 minutes. All key aspects of pain neurophysiology were explained and discussed. At the end of the first session, participants will be provided with informational handouts to support the educational process.
  Arms: MT+ PNE with MI
Other: MT — Participants in this group will be given the same MT program as "MT + PNE with MI group" without the application of PNE.
  Arms: MT
Other: Control — The participants in the control group will be provided with written instructions for performing general exercises at home. These exercises will consist of gentle stretching exercises specifically targeting the low back muscles, as well as relief positions and breathing relaxation exercises.
  Arms: Control

SUMMARY:
Non-specific chronic low back pain (NSCLBP) is characterized by persistent back pain that lasts longer than 12 weeks. This clinical trial aims to examine the short-term and long-term effects of adding Pain Neuroscience Education (PNE) with integrated Motivational Interviewing (MI) to a Manual Therapy (MT) program on pain intensity, pressure pain threshold (PPT), back performance, disability, kinesiophobia, fear and avoidance, and catastrophizing in individuals suffering from NSCLBP. The study adopts a randomized, controlled, single-blind design, with a total of 60 participants randomly allocated to three groups. The first group will receive MT and PNE with MI, the second group will receive MT alone, and the control group (third group) will follow a home-based exercise program only. All interventions will last for 4 weeks. Outcome measures will be assessed at three time points: pre-intervention, at 4 weeks, and at 6 months. The statistical analysis of the results will use a two-factor analysis of variance with repeated measurements, and the statistical significance index will be set at p < 0.05.

DETAILED DESCRIPTION:
Background: Non-specific chronic low back pain (NSCLBP) is characterized by persistent back pain that lasts longer than 12 weeks. Manual therapy (MT) is likely to exhibit short-term efficacy for NSCLBP and is recommended by clinical guidelines. Pain Neuroscience Education (PNE) is a method through which patients are taught how to alter their own pain perception using explanations, metaphors, and examples, aiming to reduce the perception of painful stimuli at the central nervous system level. Integrated Motivational Interviewing (MI) consists of a patient-centered communication approach that aims to elicit and enhance motivation for behavior change, guiding patients away from ambivalence and uncertainty.

Aim: To study the effects of adding PNE with MI to an MT program on pain, pressure pain threshold (PPT), disability, kinesiophobia, catastrophizing, fear and avoidance, and back performance in individuals suffering from NSCLBP..

Method: Sixty adults with NSCLBP will be randomly assigned into three groups of 20 people each. The first group will receive MT and PNE with integrated MI. The second group will follow MT without PNE with integrated MI. The third group (control) will receive a conventional home-based exercise program. Pain in the last 24 hours with the Numeric Pain Rating Scale (NPRS), functional ability with the Roland- Morris Disability Questionnaire (RMDQ), PPT in the lumbar region through pressure algometry, kinesiophobia with Tampa Scale for Kinesiophobia (TSK), Fear- Avoidance behavior with Fear- Avoidance Beliefs Questionnaire (FABQ), catastrophizing with Pain-Catastrophizing-Scale (PCS) and performance using the Back Performance Scale (BPS) will be evaluated at baseline, at the 4th week, and six months post-intervention..

Expected results: Manual therapy in combination with Pain Neuroscience Education have shown short term positive effects on pain, kinesiophobia and catastrophizing in individuals with non-specific low back pain. Combining Manual Therapy with Pain Neuroscience Education with integrated MI holds promise for achieving improved outcomes characterized by larger and longer-lasting effects.

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms at least 12 weeks
* Reported pain intensity of 3 or greater according to the numeric pain rating scale (NPRS)
* Written consent to participate in the study

Exclusion Criteria:

* Neuropathic pain extending along the lower limb due to nerve root compression
* Previous spine surgery
* History of spine trauma or fracture
* Cancer
* Severe osteoporosis
* Spondylo-arthropathy
* Spondylolisthesis
* Systemic inflammatory disease
* Illiterate individuals
* Diagnosed neurodegenerative diseases (e.g., Parkinson's)
* Epilepsy
* History of psychiatric disorders

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in low back pain intensity with Numeric Pain Rating Scale (NPRS) | pre-intervention, 4th week, 6-month follow-up
  This tool is an eleven-point pain scale numbered from zero to 10. The left end of the scale corresponds to zero and is marked as "No pain", whereas the right end corresponds to 10 and is marked as "Maximum pain". Consequently, a higher value indicates more intense pain. The examinee is asked to choose an integer that best reflects the intensity of their pain. The NPRS is widely used to measure pain in both clinical practice and research, showing high test-retest reliability and high conceptual construct validity.
Changes in Pressure Pain Threshold (PPT) with pressure algometry | pre-intervention, 4th week, 6-month follow-up
  Pressure pain threshold (PPT) is defined as the minimal amount of pressure that produces pain. PPT will be assessed by a digital algometer and will be evaluated bilaterally in the quadratus lumborum muscle, in the sacroiliac joints, and paravertebrally in the L4-L5 intervertebral space. The metal rod of the algometer will be placed vertically on the site and the examiner will apply gradually increasing pressure at a rate of 1Kg/s. PPT is calculated in kg/cm2 (Imamura et al., 2016).
Changes in functional capacity with the Greek Version of Roland-Morris Disability Questionnaire (RMDQ) | pre-intervention, 4th week, 6-month follow-up
  The functional ability of the participants will be evaluated with the Greek version of the Roland-Morris questionnaire, which consists of 24 questions related to daily activities that patients often report difficulty performing due to low back pain. Each positive answer earns one point and the final score is calculated by adding all the points. Therefore, the higher the score, the greater the restriction. The Greek version of the questionnaire shows satisfactory reliability and validity (ICC: 0.44-0.92) (Boscainos et al., 2003).
Changes in Kinesiophobia with Tampa Scale for Kinesiophobia (TSK) | pre-intervention, 4th week, 6-month follow-up
  The assessment of kinesiophobia will be conducted using the Tampa Scale for Kinesiophobia (TSK), a 17-item questionnaire specifically designed to evaluate fear of movement and re-injury. This scale incorporates parameters related to injury and re-injury, as well as fear-avoidance behaviors in work-related activities. Participants rate each item on a 4-point Likert-type scale, ranging from 1 (definitely disagree) to 4 (completely agree). The total score on the TSK falls within the range of 17 to 68 points, with higher scores indicating a greater level of kinesiophobia. The minimal clinically important difference (MCID) for the TSK is reported to be 8 points.
Changes in Fear- Avoidance behaviour with Fear- Avoidance Beliefs Questionnaire (FABQ) | pre-intervention, 4th week, 6-month follow-up
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a widely used assessment tool designed to measure individuals' beliefs about how physical activity and work-related activities may impact their pain and disability. It consists of fourteen items, which are scored on a 7-point Likert-type scale, ranging from "completely disagree" to "completely agree." The total score ranges from 0 to 96, with higher scores indicating stronger fear-avoidance beliefs.
Changes in Catastrophizing with Pain-Catastrophizing-Scale (PCS) | pre-intervention, 4th week, 6-month follow-up
  The Pain Catastrophizing Scale (PCS) is a widely utilized self-report questionnaire designed to assess the extent to which individuals engage in catastrophic thinking when experiencing pain. The PCS consists of 13 items, each describing different thoughts and feelings that individuals may experience when in pain. Participants rate the extent to which they experience each statement on a 5-point Likert-type scale, ranging from "not at all" to "all the time." The scale encompasses three main dimensions of catastrophizing: rumination, magnification, and helplessness.
Changes in Performance was assessed using the Back Performance Scale (BPS) | pre-intervention, 4th week, 6-month follow-up
  Performance will be assessed using the Back Performance Scale (BPS) described by Strand, Moe-Nilssen, and Ljunggren (2002). The BPS includes 5 tests of trunk mobility (sock test, pick-up test, roll-up test, fingertip-to-floor test, and lift test). Each test is scored from 0 to 3 based on the observed level of physical performance, and total score ranges from 0 to 15 points. High score indicates poor performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic Universit, Thessaloniki, Sindos Thessaloníki, Greece, Greece

IPD SHARING:
Plan to Share IPD: No